CLINICAL TRIAL: NCT03786900
Title: Fecal Microbiota Transplantation (FMT): PRIM-DJ2727
Status: Available | Type: Expanded Access
Sponsor: Herbert DuPont, MD (Other)
Responsible Party: Sponsor-Investigator, Herbert DuPont, MD, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Other Study IDs: HSC-SPH-15-0991
Record Dates: First submitted 2018-12-11; First posted 2018-12-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Clostridium Difficile Infection; Multidrug-resistant Klebsiella Pneumoniae Urinary Tract Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) product PRIM-DJ2727

SUMMARY:
The Fecal Microbiota Transplantation (FMT) product PRIM-DJ2727 is prepared from human stool from a healthy, screened donor.

Requestors will contact the study team about the product (PRIM-DJ2727) by email, visit, or phone call. A screening list for donors will be provided to make sure that the list fits the requestor's requirements. A basic fee will be requested to recover the cost of making the product. After an agreement is made, a contract will be signed between the 2 parties. A week before the treatment, requestors will contact the study team for possible FMT product delivery. Delivery method will be confirmed for delivery by personnel (within 10 minutes driving distance) or by using FedEx services. Each delivered product will have an approved delivery form signed and dated by both the person who prepared the delivery and the person who received the package.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Herbert DuPont, MD, Principal Investigator — The University of Texas Health Science Center, Houston